CLINICAL TRIAL: NCT04529187
Title: Effect of Midazolam and Dexmedetomidine on Heart Function - A Randomized MRI-based Study.
Acronym: MRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Masaryk Hospital Krajská zdravotní a.s. (Other)
Responsible Party: Principal Investigator, Nedal Omran, MD, Masaryk Hospital Krajská zdravotní a.s.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Masaryk Hospital
Record Dates: First submitted 2020-08-18; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Cardiac Function; Sedation; Magnetic Resonance Imaging
MeSH Terms: interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX group (Active Comparator): Participants allocated into this arm will undergo a baseline cardiac MRI. Then a dexmedetomidine infusion in a rate of of 0.7 ug.kg-1.hr-1will be initiated. After 5 minutes of dexmedetomidine therapy a control cardiac MRI will be performed to detect changes in heart function following sedation administration.
  Interventions: Drug: Dexmedetomidine
- MID group (Active Comparator): Participants allocated into this arm will undergo a baseline cardiac MRI. Then a single dose of midazolam (2 mg intravenously) will be given to each participant in this arm. After 5 minutes of midazolam administration a control cardiac MRI will be performed to detect changes in heart function following sedation administration.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — To monitor the changes in heart function induced after midazolam sedation using cardiac MRI.
  Other Names: Dormicum® (Roche, F. Hoffmann-La Roche Ltd Basel, Switzerland)
  Arms: MID group
Drug: Dexmedetomidine — To monitor the changes in heart function induced after dexmedetomidine sedation using cardiac MRI.
  Other Names: Dexdor® (Orion Corporation, Nasdaq OMX Helsinki: ORNAV and ORNBV, Finland)
  Arms: DEX group

SUMMARY:
To compare the changes in heart function, induced after sedation with midazolam or dexmedetomidine, using cardiac magnetic resonance imaging (MRI).

This study is a randomized unmasked study, in which participant will be allocated by the envelop method into the dexmedetomidine (DEX) group or into the midazolam (MID) group.

DETAILED DESCRIPTION:
The study will test the hypothesis that the use of dexmedetomidine leads to less negative impact on ventricular function compared to midazolam.

The study will include patients who will meet the inclusion criteria. A previous, yet unpublished, pilot study assured that a number of 15 participants in each arm is sufficient to detect statistical significant results with a statistical power of ≥ 80%. After signing the informed consent, a one-session cardiac MRI will be performed in each fasting participant before and after sedation administration (see arms and intervention). The following parameters will be recorded: end diastolic and end systolic volume, left and right ventricle stroke volume and flow velocity through the mitral valve during early and late diastole. A monitor will record values of mean blood pressure, pulse and blood oxygen saturation in 5-minute intervals.

The acquired data will be transferred to an offline workstation for postprocessing and quantification. In participants we will calculate left ventricular volumes using the well-known Simpson's formula by segmenting of endocardial borders on end-diastolic and end-systolic frames on every slice through the left ventricle.

The quantitative flow measurement will be performed using phase contrast quantification flow mapping.

Statistical analyses will be performed using STATISTICA software (data analysis software system, version 13 TIBCO Software Inc). All values will be presented as average ± standard deviation. Analysis of variance for repeated measures with post hoc Fisher's LSD test will be used for statistical testing of significant differences in each group and between the groups before and after sedation, respectively. Significance level will be accepted at α<0.05.

The participants will be monitored during sedation administration and 6 hours following sedation cessation to avoid complications that could be associated with sedation administration such as hypotension or rhythm disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were admitted due to chest pain, in whom acute coronary syndrome, pulmonary embolism and acute aortic syndrome were ruled out
* Age ≥18 and ≤ 65 years
* No contraindication to provide cardiac MRI
* No known allergy to Midazolam or Dexmedetomidine
* Signed informed consent
* No history of heart, hepatic, renal or respiratory failure

Exclusion Criteria:

* Atrial fibrilation
* Claustrophobia
* Heart Failure
* Renal Failure
* Hepatic disease
* Respiratory insufficiency
* Fertility and lactation
* Patients who cannot cooperate or refuse to sign the consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac output following sedation administration | 5 minutes following sedation administration.
  Using cardiac MRI stroke volume (measured in mL) of both heart ventricles will be registered prior and after sedation administration.
Changes in diastolic heart function following sedation administration | 5 minutes following sedation administration.
  Using cardiac MRI maximum flow velocity through the mitral valve (measured in mL/s) during early and late diastole will be measured prior and after sedation administration.

CONTACTS AND LOCATIONS:
Overall Officials: Nedal Omran, M.D, Principal Investigator — Masaryk Hospital and UJEP, Usti nad Labem, Czech Republic.
Locations (1):
- Department of Cardiology, Masaryk Hospital and UJEP, Usti nad Labem, Czech Republic., Ústí nad Labem, Czechia